CLINICAL TRIAL: NCT01446484
Title: Phase 1 Pilot Study Using Autologous CD4+CD25+FoxP3+ T Regulatory Cells and Campath-1H to Induce Renal Transplant Tolerance
Brief Title: Treatment of Children With Kidney Transplants by Injection of CD4+CD25+FoxP3+ T Cells to Prevent Organ Rejection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pirogov Russian National Research Medical University (Other)
Collaborators: Russian Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSMU-001
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: End-Stage Renal Disease; Kidney Failure
Keywords: Renal transplantation; Kidney transplantation; CD4+CD25+CD127lowFoxP3+ T Regulatory Cells; T reg; Campath
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — Cell- and Tissue-Based Therapy; Alemtuzumab; Mycophenolic Acid; Sirolimus; Tacrolimus; Cyclosporine; Everolimus; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T reg therapy (Experimental): Kidney transplantation, followed by immunotherapy given along with autologous CD4+CD25+CD127lowFoxP3+ T regulatory cells infusions
  Interventions: Biological: CD4+CD25+CD127lowFoxP3+ T regulatory cells injection; Drug: Alemtuzumab; Drug: Mycophenolate mofetil; Drug: Sirolimus; Drug: Tacrolimus; Drug: Cyclosporine; Drug: Everolimus; Procedure: Kidney transplantation
- Immunosuppression (Active Comparator): Patients will undergo immunosuppressive therapy followed by living related kidney transplantation
  Interventions: Drug: Alemtuzumab; Drug: Mycophenolate mofetil; Drug: Sirolimus; Drug: Tacrolimus; Drug: Cyclosporine; Drug: Everolimus; Procedure: Kidney transplantation

INTERVENTIONS:
Biological: CD4+CD25+CD127lowFoxP3+ T regulatory cells injection — Blood samples from patients in the experimental group will be collected twice with weekly interval in the amount of 70 ml/1,73 m2. T cells CD4+ will be separated from blood samples and frozen in liquid nitrogen. At day 30 after transplantation patients will undergo subcutaneous injection of approximately 2x 10^8 autologous T regs, expanded from previously frozen CD4+ T cells. Levels of T reg cells in patient's blood will be estimated by flow cytometry in a week after injection. That cell injection procedure will be repeated at 6 months after transplantation
  Other Names: Cell therapy
  Arms: T reg therapy
Drug: Alemtuzumab — Immunosuppressant; 2 doses of drug by intravenous infusion on Days 14 - 21 before Tx and on Day 0 after Tx
  Other Names: Campath
Drug: Mycophenolate mofetil — Immunosuppressant; oral daily dose starting Day 2-3 until withdrawal or end of the study
  Other Names: Cellcept
Drug: Sirolimus — Immunosuppressant; oral daily dose starting no earlier then after Month 1 post-transplant until withdrawal or end of the study
  Other Names: Rapamycin; Rapamune
Drug: Tacrolimus — Immunosuppressant; daily dose starting Day 0 until withdrawal or end of the study
  Other Names: Prograf
Drug: Cyclosporine — Immunosuppressant; daily dose starting Day 0 until withdrawal or end of the study
  Other Names: Neoral
Drug: Everolimus — Immunosuppressant; oral daily dose starting no earlier then after Month 1 post-transplant until withdrawal or end of the study
  Other Names: Certican; Afinitor
Procedure: Kidney transplantation — Living related kidney transplantation
  Other Names: Renal Transplantation

SUMMARY:
T regulatory cells (T regs) are responsible for immune tolerance in solid organ transplant patients. This study will evaluate the treatment of children with kidney transplants either with Campath and other immune system suppressing medications alone or in combination with injection of autologous CD4+CD25+CD127lowFoxP3+ T regulatory cells expanded ex vivo. The aim of this study is to develop a new strategy that will be more effective in preventing organ rejection and maintaining patient health.

DETAILED DESCRIPTION:
Kidney transplantation is a common procedure in hospitals, but organ rejection and serious side effects are potential problems for patients. Alemtuzumab is a monoclonal antibody to CD52 that binds to and depletes excess of T cells in the bone marrow of leukemia patients. In this study alemtuzumab will be used to deplete the recipient's white blood cells (WBCs) at the time of transplantation.

An experimental group of patients will receive two injections of autologous CD4+CD25+CD127lowFoxP3+ T regulatory cells expanded ex vivo at day 30 and day 180 after transplantation. T regulatory cells are responsible for immune system tolerance induction. Treatment with these cells is believed to create tolerance when T cell immune responses to transplant alloantigens are decreased. This study will evaluate the safety and effectiveness of an antirejection regimen including alemtuzumab and other immunosuppressive medications combined with autologous T regs injections in patients undergoing kidney transplantation (Tx). Patients will receive i.v. injection of alemtuzumab on Days 14-21 before Tx and on Day 0. Starting on Day 0, patients will begin taking either tacrolimus or cyclosporine, and on Day 2-3 - mycophenolate mofetil.

This study will continue during three years. Participants will be randomly assigned to receive either the full immunosuppressive therapy and autologous T regs by s.c. injection (group 1) or immunosuppressive therapy alone (group 2). Prior to immunosuppressive therapy in the group 1, blood samples will be collected twice with at least one-week interval between collections in the amount of 70 ml/1,73 m2 . Two ml of blood will be collected before starting of immunosuppressive therapy and levels of T regs in periphery blood will be examined by flow cytometry analysis in both groups. T cells CD4+ will be separated from these blood samples and will be frozen in liquid nitrogen.

All patients will undergo kidney transplantation. One month after transplantation the flow cytometry analysis of blood samples will be performed in both groups. The patients in group 1 will undergo by subcutaneous injection of approximately 2x10^8 autologous T regs expanded from previously frozen CD4+ cells in a month and 180 days after transplantation. One week following the injection, an additional flow cytometry analysis will be performed to evaluate T reg levels in patient's blood.

The level of T regs in patient's blood will be repeated in both groups after 90-120 days following transplantation.

Patients will be monitored during three years post-transplantation. Urine samples will be collected after one week and 1, 3, 6, and 9 months following transplantation. Kidney biopsy will be performed at Months 1, 12, and 36. Based on results of biopsy analysis, kidney function and signs of over-immunosuppression, some patients will be switched from CNIs (calcineurin inhibitors, tacrolimus or cyclosporine) to PSIs regiment (sirolimus or everolimus).

ELIGIBILITY:
Inclusion Criteria:

* Weight greater than 10 kg ( lbs)
* Will be receiving a living-related primary kidney allograft
* Negative B-cell and T-cell cytotoxic and flow cytometry crossmatch
* Normal echocardiogram (ECG) with an ejection fraction of greater than 50%
* Received full course of vaccination for hepatitis B virus (HBV), completed at least 6 weeks before transplantation, OR has naturally acquired immunity
* Parents willing to comply with the study visits

Exclusion Criteria:

* Previously received or is receiving an organ transplant other than a kidney
* Receiving an ABO incompatible donor kidney
* HIV infected
* Antibody positive for hepatitis C virus
* Surface antigen positive for HBV
* Recipient or donor is positive for tuberculosis (TB), under treatment for suspected TB, or previously exposed to TB (positive Mantoux test)
* Current cancer or a history of cancer within the 5 years prior to study entry. Patients who have had successfully treated nonmetastatic basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix are not excluded.
* Significant liver disease, defined as having continuously elevated AST (SGOT) or ALT (SGPT) levels greater than 3 times the upper value of the normal range within 28 days prior to study entry
* Uncontrolled concomitant infections, severe diarrhea, vomiting, active upper gastrointestinal tract malabsorption, active peptic ulcer, or any other unstable medical condition that could interfere with this study
* Currently receiving an investigational drug or received an investigational drug within 30 days prior to transplant
* Currently receiving any immunosuppressive agent
* Anticipated contraindication to taking medications orally or via nasogastric tube by the morning of Day 2 following completion of the transplant procedure
* Require certain medications
* Known hypersensitivity to any of the study medications,
* Any form of substance abuse, psychiatric disorder, or other condition that, in opinion of the investigator, may interfere with the study
* Anticipated contraindication to study medications administration for longer than 5 days post-transplant

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Patient and graft survival | At 1 years post-transplant

SECONDARY OUTCOMES:
Patient and graft survival | At 3 years post-transplant
Incidence rate of biopsy-proven acute rejection, defined as a renal biopsy demonstrating acute cellular or humoral rejection of Banff Grade IA or greater | 3 years
Incidence of chronic allograft nephropathy, determined using renal biopsies and laboratory values, including 24-hour urine protein excretion | 3 years
Incidence of adverse events associated with renal transplantation and immunosuppression | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana N. Bykovskaia, M.D. Ph.D., Principal Investigator — Russian State Medical University; Michael M. Kaabak, M.D. Ph.D., Principal Investigator — Boris Petrovsky's Scientific Center of Surgery Russian Academy of Medical Sciencies
Locations (2):
- Russia (2):
  - The Russian State Medical University, Moscow
  - Boris Petrovsky Scientific Center of Surgery Russian Academy of Medical Sciencies, Moscow